CLINICAL TRIAL: NCT00334607
Title: Assess the Immunogenicity of 3 Doses of Pediarix®, Prevnar® & ActHIB® Given to Healthy Infants When Administered With GSK Biologicals' 2 Dose Oral Live Attenuated Human Rotavirus Vaccine Given During the Same Vaccination Visit or Separately
Brief Title: Study of 2 Doses of HRV Vaccine Given Concomitantly or Separately With Routine Vaccinations in Healthy Infants in USA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107531
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Rotavirus
Keywords: HRV vaccine; diarrhoea; rotavirus
MeSH Terms: conditions — Rotavirus Infections; Diarrhea

INTERVENTIONS:
Biological: 2-dose oral live attenuated G1P[8] human rotavirus vaccine

SUMMARY:
The aim of this this study is to confirm absence of immune interference between HRV vaccine and routine infant vaccinations currently in use in the USA.

DETAILED DESCRIPTION:
A phase III randomized multi-center study to assess the immunogenicity of three doses of Pediarix®, Prevnar® and ActHIB® given to healthy infants at 2, 4 and 6 months of age when administered with GlaxoSmithKline (GSK) Biologicals' two-dose oral live attenuated human rotavirus (HRV) vaccine given during the same vaccination visit (at 2 and 4 months of age) or given separately (at 3 and 5 months of age).

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 -12 weeks old at Dose 1 with written informed consent.

Exclusion Criteria:

* Allergic reaction to vaccine components;
* clinically significant history of chronic GI disease (uncorrected GI congenital malformation) or other serious medical condition per investigator, received vaccines or treatment prohibited by the protocol;
* immunocompromised.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 484 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate that coadministration with HRV vaccine does not impair the immune response to all antigens contained in each of the routine infant vaccines.

SECONDARY OUTCOMES:
Assess immunogenicity and safety of HRV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (40):
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Cabot, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Commerce Twp, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Bryson City, North Carolina
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Deerfield, North Carolina
  - GSK Investigational Site, Franklin, North Carolina
  - GSK Investigational Site, Laurinburg, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dennehy PH, Bertrand HR, Silas PE, Damaso S, Friedland LR, Abu-Elyazeed R. Coadministration of RIX4414 oral human rotavirus vaccine does not impact the immune response to antigens contained in routine infant vaccines in the United States. Pediatrics. 2008 Nov;122(5):e1062-6. doi: 10.1542/peds.2008-1059. PMID 18977955
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107531 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register